CLINICAL TRIAL: NCT01798407
Title: A Clinical Pilot Study Examining Bilateral Inhibition of the Lateral Habenula as a Target for Deep Brain Stimulation in Intractable Depression
Brief Title: DBS of the Lateral Habenula in Treatment-Resistant Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne Goodman MD (Other)
Responsible Party: Sponsor-Investigator, Wayne Goodman MD, Principal Investigator; Chairman, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H40307; 49593 (Other: BCM); 277909 (Other: Simons Foundation); HSM#12-00467 (Other Grant/Funding Number: MSSM IRB); GCO 12-1815 (Other: MSSM IRB)
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Treatment Resistant Major Depressive Disorder
Keywords: Deep Brain Stimulation; Major Depressive Disorder; Depression; Lateral Habenula; Intractable Depression; Treatment Resistant Depression (TRD)
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder, Treatment-Resistant | interventions — Deep Brain Stimulation; Random Allocation

STUDY DESIGN:
Intervention Model Description: all subjects will receive bilateral surgical implantation of DBS system. Those who respond at 12 months will enter a randomized, staggered withdrawal phase. See masking description below.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During staggered withdrawal phase, double blind discontinuation will be attempted on either the 12 or 13 month visit. Stimulation intensity will be decreased by 50% and then completely discontinued two weeks later. Subjects will be seen every 2 weeks until 15 months post activation or escape criteria are met. These escape criteria include relapse at 2 visits, hospitalization, active suicidal ideation, or withdrawing consent. If any of these criteria are met, the blind will be broken and open treatment will be resumed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Activa Tremor Control Sys (DBS Implant) (Experimental): all subjects will receive bilateral surgical implantation of DBS system. Those who respond at 12 months will enter a randomized, staggered withdrawal phase.
  Interventions: Device: Activa Tremor Control Sys (DBS Implant)
- Randomized, staggered withdrawal phase (Experimental): For responders only: double blind discontinuation will be attempted on either the 12 or 13 month visit. Stimulation intensity will be decreased by 50% and then completely discontinued two weeks later. Subjects will be seen biweekly until 15 months post activation or escape criteria are met. These escape criteria include relapse at 2 visits, hospitalization, active suicidal ideation, or withdrawing consent. If any of these criteria are met, the blind will be broken and open treatment will be resumed.
  Interventions: Other: Randomized, staggered withdrawal phase

INTERVENTIONS:
Device: Activa Tremor Control Sys (DBS Implant) — DBS system consists of the Activa RC 37612 System (Implantable Pulse Generator with Model 37085 Extensions (40 to 95cm), Activa Patient Programmer, and Medtronic Model 3389 DBS Lead). This system is commercially approved for the treatment of chronic, intractable Parkinson's Disease. It will be used with the Model SP-10344 Memory Mod Software which enables the physician to program the Implantable Pulse Generator to a higher frequency.
  Other Names: Deep Brain Stimulation System; DBS; Activa RC System
  Arms: Activa Tremor Control Sys (DBS Implant)
Other: Randomized, staggered withdrawal phase — For responders only: double blind discontinuation will be attempted on either the 12 or 13 month visit. Stimulation intensity will be decreased by 50% and then completely discontinued two weeks later. Subjects will be seen biweekly until 15 months post activation or escape criteria are met. These escape criteria include relapse at 2 visits, hospitalization, active suicidal ideation, or withdrawing consent. If any of these criteria are met, the blind will be broken and open treatment will be resumed.
  Arms: Randomized, staggered withdrawal phase

SUMMARY:
This research study will investigate the safety, tolerability, and benefit of bilateral deep brain stimulation (DBS) to the lateral habenula in subjects with treatment-resistant major depression (TRD) secondary to either nonpsychotic unipolar major depressive disorder (MDD), or bipolar disorder (BD) I. Six adult subjects with TRD will be treated in this single-site study at Baylor College of Medicine; subjects will be chronically symptomatic with significant functional disability, and will have demonstrated resistance to standard somatic and pharmacotherapeutic treatments. The primary outcome measure will be the change in the 17-item Hamilton Depression Rating Scale (HDRS^17) six months after the commencement of stimulation.

DETAILED DESCRIPTION:
This research study includes the following parts: 1. medical, psychiatric, and cognitive evaluations 2. implantation of the brain stimulation system, and 3. follow up including programming and psychiatric testing after the implantation

1. Medical, psychiatric, and cognitive evaluations:

   For those subjects that are found to be eligible and agree to participate in the study, they will be asked more detailed questions about their symptoms, mood, and thinking on another visit before receiving the implantation. The investigator will ask detailed questions about the subject's psychiatric and medical history, and will ask for a list of medications along with response to previous treatments. The subject will also be asked to fill out several questionnaires.

   Subjects will be asked to give a sample of both blood and urine for standard lab evaluations. All subjects will be tested for the presence of drugs of abuse in their urine. All women of child bearing potential will also be tested for pregnancy. If any of the test results are positive, the subject cannot continue to be part of this study, but can receive other standard clinical care by a treating psychiatrist.

   As part of the pre-operative clinical evaluation, all subjects will be evaluated by a neurosurgeon, and, potentially, a medical specialist for surgical optimization, as well as an anesthesiologist for an intra-operative risk assessment. Prior to surgery, an independent evaluator who is not affiliated with the research study will confirm the diagnosis of MDD and assess the subject's understanding of the risks of the surgery and follow-up care.

   Additionally, subjects will have two pre-surgical magnetic resonance imaging (MRI) scans. This is to ensure accurate placement of the system leads and will take place the the month before surgery. Subjects will also have neuropsychological testing (cognitive tests of memory and thinking skills) before and after surgery.
2. Implantation of the brain stimulation system:

The brain stimulation system is implanted inside the subject's body. The implanted system is made up of three major parts:

* The leads are made of four insulated wires with four electrodes at the end.
* The extensions connect the lead to the neurostimulator (power source).
* The neurostimulator (battery) is the power source of the system.

The neurostimulator is a metal "can", which depending on the model the subject receives, will be in the range of about 2 or 3 inches in diameter and about ½ inch thick. It contains a small battery and produces the electrical impulses needed for stimulation. For this study a rechargeable battery will be used; this battery cannot be replaced without replacing the entire neurostimulator. Replacing the neurostimulator involves minor surgery. Although battery life varies for each subject depending on the type and intensity of stimulation needed for good symptom relief, the use of a rechargeable battery will extend the time before it must be replaced. A hand held control magnet is used to turn the therapy on and off.

Subjects will have two leads and one neurostimulator implanted,. The surgeon may place the neurostimulator either near the collarbone or within the abdomen.

Devices will be implanted in a staged fashion, meaning that subjects will have each lead placed in one individual procedure. The lead extensions and neurostimulator will be placed during the second procedure, after the second lead has been placed. The lead implant surgeries will take place approximately 1-2 weeks apart. On the evenings before surgeries, subjects may be instructed to stop taking all of their medications. This is so the effect of the deep brain stimulation on the subject's symptoms can best be determined. Subjects will be admitted to the hospital the mornings of each surgery and may have their head shaved prior to surgery to help prevent infection. Additionally, the surgical team will assess the subject's emotional and physical status on the morning of the second surgery and will notify the study team if there are any concerns.

The day of each surgery, the following steps may occur:

1. Pictures of the brain will be taken using computer-aided tomography (CT) scans and 3D imaging. This will be combined with the previous MRI scans and allow the surgeon to determine the area in the brain where the leads will be placed. A CT scan - also called CT or computerized tomography - is an X-ray procedure where a high-speed computer is used to make multiple images or pictures of the body. Subjects will be asked to lie still on a table and at time may have to hold their breath for a few seconds in order to avoid blurring the pictures. Subjects may have 1 CT scan before and after each surgery to ensure the leads are in the correct locations on the brain.
2. In the operating room, a metal frame will be attached to the head. The frame is a special instrument that allows the surgeon to find the correct path to the target site in the brain. Local anesthetic will be given so that the pins, which hold the frame to the head, do not hurt.
3. Subjects will be positioned on the operating table and a catheter will be inserted and antibiotics will be given through an intravenous (IV) line placed in the arm. Vital signs will be monitored. The metal frame attached to the subject's head will also be attached to the operating table for safety. The subject's head will be sterile prepared for the procedure.
4. A small hole will be drilled in the skull, for the lead to be implanted that day (2 total leads placed 1 at a time on 2 separate surgery days). The subject will receive local anesthesia before this procedure.
5. The lead is then passed into the brain to the desired site. Test stimulation will be performed to determine if there are unwanted side effects. Once test stimulation is complete, the device will be turned "off" until the entire system has been implanted (i.e., both leads, extensions, and neurostimulator) and the subject has recovered from the surgeries.
6. A cap will be placed over the hole in the skull. The cap also holds the lead in position.
7. The metal frame is then removed from the subject's head.
8. After the implantation procedures, additional CT brain imaging will be performed.
9. The extensions and neurostimulator will be placed during the second surgery (about two weeks following the first surgery), after the second lead has been placed on the other side of the brain. This part is performed under general anesthesia. Some additional blood tests may be performed to confirm the subject is stable.

The subject will be admitted the morning of surgery and stay in the hospital overnight after each surgery. They will typically be discharged the next day once it is determined that they are in stable condition

Interim Clinical Assessment: If the second surgery is to be performed within 2 weeks of the first surgery, the subject may not have an interim clinical assessment performed. However, if your second stage surgery is scheduled 2 weeks or more after the first stage, this visit will be performed. During this visit, the subject will be evaluated on recovery from the first surgery and asked about depressive symptoms. Subjects will also be asked to fill out several questionnaires. This visit will take place at the Baylor Psychiatry Clinic and will last approximately one hour.

Either way, for both surgeries, standard surgical follow up procedures will be followed. The surgical team will follow up with the subject after each surgery on the day they have surgery and prior to discharge while they are still in the hospital. The surgical team will also follow up with the subject within a week of discharge. They will assess the subject's emotional and physical status and will bring the subject in as soon as possible for further evaluation if there are any concerns.

3) Follow-up programming and psychiatric assessments The study physician see subjects for follow up after surgery. Follow up visits are scheduled after subjects are implanted. During these visits, the study physicians or other clinicians will assess the subject's condition using various standardized questionnaires.

Frequent, non-invasive adjustment to the stimulation parameters may be required to achieve optimal symptom response. This adjustment period may take weeks or months.

The DBS device will be turned "on" during the first programming visit with the study doctor, about 2 weeks after the second surgery.

4) Duration of treatment The optimization period generally lasts about 8 weeks, after which modulation appointments are scheduled monthly or on an as needed basis. A CT scan will be performed at Month 3 to check on the placement of the subject's leads. The subject will receive up to 5 total CT scans. 1 CT scan before and after each surgery and 1 CT scan at the 3-month checkup mark. These 5 CT scans are to ensure the leads are in the correct locations of the subject's brain. If a subject responds to the treatment, stimulation may be temporarily discontinued between months 12 and 18 to find out if the response is because of the treatment. The subject will not be told when this discontinuation occurs and they will be carefully monitored during this time (seen approximately every 2 weeks). If symptoms worsen, the subject will be informed if stimulation was discontinued, and they will have the option to have stimulation restarted. If the subject continues to do well without stimulation, they may be offered the opportunity to continue without stimulation, consider removing the device, or to restart stimulation.

For subjects that do not respond to the DBS treatment, the system will remain implanted unless the subject desires for it to be removed or it is medically necessary that it be removed. After the End of the Study (Month 18), the device will remain implanted in subjects that are doing well clinically.

Because the battery life is approximately 7-9 years, every 7-9 years batteries will need to be replaced. This requires subjects to undergo a brief surgery to have the neurostimulator replaced - the neurostimulator contains a small rechargeable battery and produces the electrical impulses needed for stimulation. When the battery can no longer be recharged, the neurostimulator must be replaced. Once a subject has exited the study, their insurance may not pay for device replacements or other medical care related to the device.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (non-pregnant) between ages 21 and 70;
* DSM-5 diagnosis (assessed by Structured Clinical Interview for DSM-5, SCID-5) of a current major depressive episode (MDE), recurrent or single episode with first episode before age 45, secondary to either nonpsychotic unipolar major depressive disorder (MDD)or bipolar disorder (BD) I;
* Chronic illness with current MDE ≥ 24 months duration and/or recurrent illness with at least a total of 4 lifetime episodes (including current episode ≥ 12 months);
* For subjects with a bipolar disorder: the last manic or hypomanic episode must have been ≥ 24 months before study enrollment and patients must be maintained on a mood stabilizer (e.g. lithium or another mood stabilizer approved for bipolar disorder).
* Treatment resistance (defined by criteria on the Antidepressant Treatment History Form): Failure (i.e. persistence of the major depressive episode) to respond to a minimum of three adequate depression treatments from at least two different treatment categories (e.g. SSRI's, TCA's, other antidepressants, lithium-addition, irreversible MAO-inhibitor, antidepressant augmentation with an atypical antipsychotic medication); also, if diagnosed as bipolar, failure to respond to (or inability to tolerate) a minimum of three treatments approved for bipolar disorder, including lithium and at least one medication FDA-approved for bipolar depression (e.g., olanzapine/fluoxetine combination, quetiapine, lurasidone).
* Previous trial of ECT (lifetime)
* Symptom Severity: HDRS17 ≥ 21; on two separate assessments (at initial screening and 1 week before surgery), over a 1-month period;
* Normal brain MRI within 3 months of surgery;
* Stable antidepressant medical regimen for the month preceding surgery
* Modified mini-mental state examination (MMSE) score ≥ 27;
* Normal thyroid stimulating hormone (TSH) level within 12 months of study entry;
* Other medical conditions must be stable for at least 1 year;
* Anticipates a stable psychotropic medication regimen in the next 24 months;
* Subject must be able to identify a family member, physician, or friend who will participate in the Treatment Contract;
* Able and willing to give informed consent.

Exclusion Criteria:

* Schizophrenia Spectrum or Other Psychotic Disorders (excluding Schizotypal (Personality) Disorder and Substance/Medication Induced Psychotic Disorder); presence of primary or serious (requiring additional treatment) disorders: comorbid obsessive compulsive disorder, post-traumatic stress disorder, panic disorder, bulimia or anorexia, in the last year;
* Cluster A or B personality disorder;
* Alcohol or substance abuse/dependence within 6 months, excluding nicotine and cannabis provided that participant either a) has a legal prescription or b) is a legal resident of a state where recreational cannabis use is legal;
* Current substantial suicidal risk as defined by a plan or clear immediate intent for self-harm, or had a serious suicide attempt within the last year;
* Neurological disease that impairs motor, sensory or cognitive function or that requires intermittent or chronic medication (e.g., Parkinson's disease, MS, stroke);
* Any history of seizure disorder or hemorrhagic stroke;
* Any medical contraindication to surgery, including infection or coagulopathy;
* Participation in another drug, device, or biological trial within 30 days;
* Current implanted stimulation devices including cardiac pacemakers, defibrillators, and neurostimulators including spinal cord stimulators, and deep brain stimulators;
* Does not have adequate family/friend support as determined by psychological screening and/or interview;
* Abnormal brain MRI;
* Unable to maintain a stable psychotropic medication regimen in the next 24 months
* Pregnant or has plans to become pregnant in the next 24 months.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in HDRS^17 score from baseline to 6 months after the commencement of stimulation | baseline, Month 6, Month 12 and 18 months
  'Response' is categorically defined as a ≥ 50% reduction in the HDRS17 score relative to the baseline assessment. 'Remission' is defined as an absolute HDRS17 score < 8. Study success criteria will be defined as ≥ 3 of the 6 patients meeting the individual subject success criteria of response or remission by HDRS17 score at the 6 month time point.

SECONDARY OUTCOMES:
MADRS (Montgomery and Asberg Depression Rating Scale) | baseline, Month 6, Month 12 and 18 months
  Clinician administered evaluation of depressive symptoms
Clinical Global Impression of Severity (CGI-S) | baseline, Month 6, Month 12 and 18 months
  Clinician Administered assessment
Clinical Global Impression of Improvement (CGI-I) | baseline, Month 6, Month 12 and 18 months
  Clinician administered assessment
Young Mania Rating Scale (YMRS) | baseline, Month 6, Month 12 and 18 months
  Clinician administered assessment
Columbia Suicide Severity Rating Scale (C-SSRS) | baseline, Month 6, Month 12 and 18 months
  Clinician administered assessment
Neuropsychological Battery | baseline, Month 6, Month 12 and 18 months
  Clinician administered assessment includes WAIS-IV subscales subscales: Digit Span, Information, Coding, Similarities, and Visual Puzzles; TMT (Trail Making Tests) A and B; Neuropsychological Assessment Battery (NAB): Naming Test; JLO, (Benton Judgment of Line Orientation Test [Forms H and V]); HVLT-R (Hopkins Verbal Learning Test-R [Forms 1, 2, 3, and 4]); BVMT-R (Brief Visual Spatial Memory Test, Revised [Forms 1, 2, 3, and 4]); GPT (Grooved Pegboard Test); COWAT (Controlled Oral Word Association Test) with semantic fluency; WCST (Wisconsin Card Sorting Test) - short version (64 item); Stroop (Stroop Color Word Test); IGT(Iowa Gambling Task)
QIDS-SR (Quick Inventory of Depressive Symptomatology) | baseline, Month 6, Month 12 and 18 months
  Subject self rated assessment
Generalized Anxiety Disorder 7-item Scale (GAD-7) | baseline, Month 6, Month 12 and 18 months
  Subject self rated assessment
Sheehan Disability Scale | baseline, Month 6, Month 12 and 18 months
  Subject self rated assessment
PRISE (The Patient Rated Inventory of Side Effects) | baseline, Month 6, Month 12 and 18 months
  Subject self report of adverse events (and collection)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne K Goodman, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bewernick BH, Hurlemann R, Matusch A, Kayser S, Grubert C, Hadrysiewicz B, Axmacher N, Lemke M, Cooper-Mahkorn D, Cohen MX, Brockmann H, Lenartz D, Sturm V, Schlaepfer TE. Nucleus accumbens deep brain stimulation decreases ratings of depression and anxiety in treatment-resistant depression. Biol Psychiatry. 2010 Jan 15;67(2):110-6. doi: 10.1016/j.biopsych.2009.09.013. PMID 19914605
- [Background] Kennedy SH, Giacobbe P, Rizvi SJ, Placenza FM, Nishikawa Y, Mayberg HS, Lozano AM. Deep brain stimulation for treatment-resistant depression: follow-up after 3 to 6 years. Am J Psychiatry. 2011 May;168(5):502-10. doi: 10.1176/appi.ajp.2010.10081187. Epub 2011 Feb 1. PMID 21285143
- [Background] Lozano AM, Mayberg HS, Giacobbe P, Hamani C, Craddock RC, Kennedy SH. Subcallosal cingulate gyrus deep brain stimulation for treatment-resistant depression. Biol Psychiatry. 2008 Sep 15;64(6):461-7. doi: 10.1016/j.biopsych.2008.05.034. Epub 2008 Jul 18. PMID 18639234
- [Background] Malone DA Jr, Dougherty DD, Rezai AR, Carpenter LL, Friehs GM, Eskandar EN, Rauch SL, Rasmussen SA, Machado AG, Kubu CS, Tyrka AR, Price LH, Stypulkowski PH, Giftakis JE, Rise MT, Malloy PF, Salloway SP, Greenberg BD. Deep brain stimulation of the ventral capsule/ventral striatum for treatment-resistant depression. Biol Psychiatry. 2009 Feb 15;65(4):267-75. doi: 10.1016/j.biopsych.2008.08.029. Epub 2008 Oct 8. PMID 18842257
- [Background] Mayberg HS, Lozano AM, Voon V, McNeely HE, Seminowicz D, Hamani C, Schwalb JM, Kennedy SH. Deep brain stimulation for treatment-resistant depression. Neuron. 2005 Mar 3;45(5):651-60. doi: 10.1016/j.neuron.2005.02.014. PMID 15748841
- [Background] Sartorius A, Kiening KL, Kirsch P, von Gall CC, Haberkorn U, Unterberg AW, Henn FA, Meyer-Lindenberg A. Remission of major depression under deep brain stimulation of the lateral habenula in a therapy-refractory patient. Biol Psychiatry. 2010 Jan 15;67(2):e9-e11. doi: 10.1016/j.biopsych.2009.08.027. No abstract available. PMID 19846068
- [Background] Schlaepfer TE, Cohen MX, Frick C, Kosel M, Brodesser D, Axmacher N, Joe AY, Kreft M, Lenartz D, Sturm V. Deep brain stimulation to reward circuitry alleviates anhedonia in refractory major depression. Neuropsychopharmacology. 2008 Jan;33(2):368-77. doi: 10.1038/sj.npp.1301408. Epub 2007 Apr 11. PMID 17429407
- [Background] Bewernick BH, Kayser S, Sturm V, Schlaepfer TE. Long-term effects of nucleus accumbens deep brain stimulation in treatment-resistant depression: evidence for sustained efficacy. Neuropsychopharmacology. 2012 Aug;37(9):1975-85. doi: 10.1038/npp.2012.44. Epub 2012 Apr 4. PMID 22473055
- [Background] Binder DK, Rau G, Starr PA. Hemorrhagic complications of microelectrode-guided deep brain stimulation. Stereotact Funct Neurosurg. 2003;80(1-4):28-31. doi: 10.1159/000075156. PMID 14745205
- [Background] Dougherty DD, Rezai AR, Carpenter LL, Howland RH, Bhati MT, O'Reardon JP, Eskandar EN, Baltuch GH, Machado AD, Kondziolka D, Cusin C, Evans KC, Price LH, Jacobs K, Pandya M, Denko T, Tyrka AR, Brelje T, Deckersbach T, Kubu C, Malone DA Jr. A Randomized Sham-Controlled Trial of Deep Brain Stimulation of the Ventral Capsule/Ventral Striatum for Chronic Treatment-Resistant Depression. Biol Psychiatry. 2015 Aug 15;78(4):240-8. doi: 10.1016/j.biopsych.2014.11.023. Epub 2014 Dec 13. PMID 25726497
- [Background] Ely BA, Xu J, Goodman WK, Lapidus KA, Gabbay V, Stern ER. Resting-state functional connectivity of the human habenula in healthy individuals: Associations with subclinical depression. Hum Brain Mapp. 2016 Jul;37(7):2369-84. doi: 10.1002/hbm.23179. Epub 2016 Mar 16. PMID 26991474
- [Background] Fenoy AJ, Simpson RK Jr. Risks of common complications in deep brain stimulation surgery: management and avoidance. J Neurosurg. 2014 Jan;120(1):132-9. doi: 10.3171/2013.10.JNS131225. Epub 2013 Nov 15. PMID 24236657
- [Background] Holtzheimer PE, Kelley ME, Gross RE, Filkowski MM, Garlow SJ, Barrocas A, Wint D, Craighead MC, Kozarsky J, Chismar R, Moreines JL, Mewes K, Posse PR, Gutman DA, Mayberg HS. Subcallosal cingulate deep brain stimulation for treatment-resistant unipolar and bipolar depression. Arch Gen Psychiatry. 2012 Feb;69(2):150-8. doi: 10.1001/archgenpsychiatry.2011.1456. Epub 2012 Jan 2. PMID 22213770
- [Background] Holtzheimer PE, Husain MM, Lisanby SH, Taylor SF, Whitworth LA, McClintock S, Slavin KV, Berman J, McKhann GM, Patil PG, Rittberg BR, Abosch A, Pandurangi AK, Holloway KL, Lam RW, Honey CR, Neimat JS, Henderson JM, DeBattista C, Rothschild AJ, Pilitsis JG, Espinoza RT, Petrides G, Mogilner AY, Matthews K, Peichel D, Gross RE, Hamani C, Lozano AM, Mayberg HS. Subcallosal cingulate deep brain stimulation for treatment-resistant depression: a multisite, randomised, sham-controlled trial. Lancet Psychiatry. 2017 Nov;4(11):839-849. doi: 10.1016/S2215-0366(17)30371-1. Epub 2017 Oct 4. PMID 28988904
- [Background] Jimenez F, Velasco F, Salin-Pascual R, Hernandez JA, Velasco M, Criales JL, Nicolini H. A patient with a resistant major depression disorder treated with deep brain stimulation in the inferior thalamic peduncle. Neurosurgery. 2005 Sep;57(3):585-93; discussion 585-93. doi: 10.1227/01.neu.0000170434.44335.19. PMID 16145540
- [Background] Kiening K, Sartorius A. A new translational target for deep brain stimulation to treat depression. EMBO Mol Med. 2013 Aug;5(8):1151-3. doi: 10.1002/emmm.201302947. Epub 2013 Jul 4. No abstract available. PMID 23828711
- [Background] Kim JW, Naidich TP, Ely BA, Yacoub E, De Martino F, Fowkes ME, Goodman WK, Xu J. Human habenula segmentation using myelin content. Neuroimage. 2016 Apr 15;130:145-156. doi: 10.1016/j.neuroimage.2016.01.048. Epub 2016 Jan 27. PMID 26826517
- [Background] Kubu CS, Malone DA, Chelune G, Malloy P, Rezai AR, Frazier T, Machado A, Rasmussen S, Friehs G, Greenberg BD. Neuropsychological outcome after deep brain stimulation in the ventral capsule/ventral striatum for highly refractory obsessive-compulsive disorder or major depression. Stereotact Funct Neurosurg. 2013;91(6):374-8. doi: 10.1159/000348321. Epub 2013 Oct 9. PMID 24108099
- [Background] Liu JK, Soliman H, Machado A, Deogaonkar M, Rezai AR. Intracranial hemorrhage after removal of deep brain stimulation electrodes. J Neurosurg. 2012 Mar;116(3):525-8. doi: 10.3171/2011.10.JNS11465. Epub 2011 Dec 2. PMID 22136644
- [Background] Lozano AM, Giacobbe P, Hamani C, Rizvi SJ, Kennedy SH, Kolivakis TT, Debonnel G, Sadikot AF, Lam RW, Howard AK, Ilcewicz-Klimek M, Honey CR, Mayberg HS. A multicenter pilot study of subcallosal cingulate area deep brain stimulation for treatment-resistant depression. J Neurosurg. 2012 Feb;116(2):315-22. doi: 10.3171/2011.10.JNS102122. Epub 2011 Nov 18. PMID 22098195
- [Background] Lujan JL, Chaturvedi A, Choi KS, Holtzheimer PE, Gross RE, Mayberg HS, McIntyre CC. Tractography-activation models applied to subcallosal cingulate deep brain stimulation. Brain Stimul. 2013 Sep;6(5):737-9. doi: 10.1016/j.brs.2013.03.008. Epub 2013 Apr 6. PMID 23602025
- [Background] Merkl A, Schneider GH, Schonecker T, Aust S, Kuhl KP, Kupsch A, Kuhn AA, Bajbouj M. Antidepressant effects after short-term and chronic stimulation of the subgenual cingulate gyrus in treatment-resistant depression. Exp Neurol. 2013 Nov;249:160-8. doi: 10.1016/j.expneurol.2013.08.017. Epub 2013 Sep 5. PMID 24012926
- [Background] Neimat JS, Hamani C, Giacobbe P, Merskey H, Kennedy SH, Mayberg HS, Lozano AM. Neural stimulation successfully treats depression in patients with prior ablative cingulotomy. Am J Psychiatry. 2008 Jun;165(6):687-93. doi: 10.1176/appi.ajp.2008.07081298. No abstract available. PMID 18519534
- [Background] Neumann WJ, Huebl J, Brucke C, Gabriels L, Bajbouj M, Merkl A, Schneider GH, Nuttin B, Brown P, Kuhn AA. Different patterns of local field potentials from limbic DBS targets in patients with major depressive and obsessive compulsive disorder. Mol Psychiatry. 2014 Nov;19(11):1186-92. doi: 10.1038/mp.2014.2. Epub 2014 Feb 11. PMID 24514569
- [Background] Perez-Caballero L, Perez-Egea R, Romero-Grimaldi C, Puigdemont D, Molet J, Caso JR, Mico JA, Perez V, Leza JC, Berrocoso E. Early responses to deep brain stimulation in depression are modulated by anti-inflammatory drugs. Mol Psychiatry. 2014 May;19(5):607-14. doi: 10.1038/mp.2013.63. Epub 2013 May 28. PMID 23711979
- [Background] Puigdemont D, Portella M, Perez-Egea R, Molet J, Gironell A, de Diego-Adelino J, Martin A, Rodriguez R, Alvarez E, Artigas F, Perez V. A randomized double-blind crossover trial of deep brain stimulation of the subcallosal cingulate gyrus in patients with treatment-resistant depression: a pilot study of relapse prevention. J Psychiatry Neurosci. 2015 Jul;40(4):224-31. doi: 10.1503/jpn.130295. PMID 25652752
- [Background] Ramasubbu R, Anderson S, Haffenden A, Chavda S, Kiss ZH. Double-blind optimization of subcallosal cingulate deep brain stimulation for treatment-resistant depression: a pilot study. J Psychiatry Neurosci. 2013 Sep;38(5):325-32. doi: 10.1503/jpn.120160. PMID 23527884
- [Background] Riva-Posse P, Choi KS, Holtzheimer PE, McIntyre CC, Gross RE, Chaturvedi A, Crowell AL, Garlow SJ, Rajendra JK, Mayberg HS. Defining critical white matter pathways mediating successful subcallosal cingulate deep brain stimulation for treatment-resistant depression. Biol Psychiatry. 2014 Dec 15;76(12):963-9. doi: 10.1016/j.biopsych.2014.03.029. Epub 2014 Apr 13. PMID 24832866
- [Background] Schlaepfer TE, Bewernick BH, Kayser S, Madler B, Coenen VA. Rapid effects of deep brain stimulation for treatment-resistant major depression. Biol Psychiatry. 2013 Jun 15;73(12):1204-12. doi: 10.1016/j.biopsych.2013.01.034. Epub 2013 Apr 3. PMID 23562618